CLINICAL TRIAL: NCT06552507
Title: The Outcome of Injured Cervical Spinal Cord with Uncontrolled Swelling Under Duraplasty
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2312250059
Record Dates: First submitted 2024-07-16; First posted 2024-08-14 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-05

CONDITIONS: Spine Injury; Cord Injury, Spinal; Cord Infarction Spinal; Incomplete Spinal Cord Injury; Complete Spinal Cord Injury
Keywords: Duroplasty; spinal cord injury; Dura augmentation
MeSH Terms: conditions — Spinal Injuries; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Laminectomy with Duroplasty (Experimental): Duroplasty
  Interventions: Procedure: Duroplasty
- Laminectomy only (No Intervention): laminectomy without duroplasty

INTERVENTIONS:
Procedure: Duroplasty — The investigators open the dura from midline and repaired with fish mouth for dura augmentation
  Arms: Laminectomy with Duroplasty

SUMMARY:
Overall Objective: To assess whether incorporating duraplasty alongside bony decompression enhances motor function outcomes in individuals following Traumatic Spinal Cord Injury (TSCI).

Rationale for Research:

In a systematic review, individuals suffering from cervical Traumatic Spinal Cord Injuries (TSCIs) identified specific priorities for improvement in their quality of life. These priorities encompassed enhanced arm and hand function, improved bladder and bowel control, sexual function, and the nurturing of personal relationships with their families and friends.

In this context, the investigators posit that augmenting standard treatment with expansion duraplasty has the potential to address several critical aspects of TSCI. Our hypothesis centers on the idea that the incorporation of duraplasty into the treatment regimen can lead to a reduction in spinal cord compression, an enhancement in Spinal Cord Perfusion Pressure (SCPP), an amelioration in spinal cord metabolism, and a mitigation of inflammation at the injury site. The investigatorsanticipate that these physiological and metabolic enhancements will contribute to increased neuronal survival, ultimately resulting in improved motor outcomes. These improved motor outcomes, in turn, are expected to translate into enhanced limb function, superior bladder and bowel control, and an overall improvement in the quality of life for the patients.

Our investigative focus encompasses a comprehensive examination of the impact of duraplasty on various facets of spinal cord physiology, metabolism, inflammation, motor and sensory performance, and Health-Related Quality of Life (HRQoL) measures. These HRQoL measures encompass aspects such as hand function, ambulation, bladder and bowel function, as well as the mental, emotional, and social well-being of the patients.

In the north area of R.O.C, individuals with TSCI are initially admitted to Linkou Chang Guan Memorial Hospital, where they typically undergo surgery involving spinal instrumentation (e.g., screws and rods) to address deformities and instability. Bony decompression, typically carried out through laminectomy, is a common surgical intervention aimed at addressing the adverse effects of bony compression on the spinal cord. It is worth noting that a significant majority of surgeons (ranging from 85% to 96%) advocate for bony decompression as a primary treatment for TSCI, as recommended by the National Institute for Health and Care Excellence (NICE) guidelines in 2016. However, the effectiveness of bony decompression in improving outcomes following TSCI remains a topic of debate and uncertainty, largely due to the absence of robust evidence from randomized controlled trials (RCTs).

Our proposal suggests that bony decompression in isolation may offer only partial relief to the swollen and injured spinal cord, which continues to experience compression against the dura. This may explain the persisting uncertainty surrounding the benefits of bony decompression in TSCI treatment. Achieving adequate cord decompression through surgical intervention assumes particular importance in this context, given the lack of pharmaceutical treatments proven to enhance outcomes in individuals with acute and severe TSCI. While the administration of methylprednisolone initially showed promise, subsequent trials, observational studies, and meta-analyses have cast doubt on its efficacy and raised concerns about potential harm.

The management of TSCI in the R.O.C is characterized by considerable variation among major trauma centers, encompassing diverse practices related to factors such as target blood pressure, choice of anesthetic agents, extent of monitoring (including the use of arterial and central lines), and timing of surgery. To circumvent these controversies and differences in practice, the "The outcome of Injured cervical Spinal Cord with Uncontrolled Swelling under Duraplasty" trial has been meticulously designed in a single major trauma center to allow participating surgeon can follow the same protocol about time to surgery and medically management.

The "The outcome of Injured cervical Spinal Cord with Uncontrolled Swelling under Duraplasty" trial was conceived with the aim of addressing these critical questions surrounding TSCI management, ultimately seeking to improve the outcomes and quality of life for individuals grappling with this challenging condition.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Severe cervical (C2 - T1) traumatic spinal cord injury (AIS grade A-C)
* Deemed to require and be suitable for surgery that includes laminectomy or diskectomy by local surgeon
* Surgery within 72 hours of traumatic spinal cord injury
* Able to provide informed consent or consultee declaration or proxy consent

Exclusion Criteria:

* Life-limiting or rehabilitation-restricting co-morbidities
* Thoracic or lumbar traumatic spinal cord injury
* Probable dural tear due to injury
* Other central nervous system disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Delta-AMS | 6 months post-randomisation minus pre-operative baseline
  The change in American Spinal Injury Association Impairment Scale (AIS) motor score. We also call it Delta-AMS, and the maximum is 100 and the minimum is 0. If the Delta-AMS is higher then it mean the patient has better recovery of the muscle power regained and vice versa.

SECONDARY OUTCOMES:
CUE-Q | 3, 6 and 12 month
  Capabilities of Upper Extremity Test (CUE-Q) [Maximum= 128, Minimum: 0, Higher the better]
WISCI-II | 3, 6 and 12 month
  Walking Index for Spinal Cord Injury (WISCI-II) [Level 0--20, the higher level the better outcome]
SCIM-II | 3, 6 and 12 month
  Spinal Cord Independence Measure (SCIM-II) [Maximum: 100, Minimum:0, the higher score the better outcome] [weight in kilograms, height in meters]
SF-36 | 3, 6 and 12 months.
  life quality the evaluation scale is not the simple meaning of score, there are eight category of the scale, and each has it's specific score sum of the scale .
  for example the [Physical functioning, PF] is the sum of the question 3, and the maximum and minimum are 30 and 10 respectively.

REFERENCES:
- [Background] van Daalen Wetters T, Coffino P. Cultured S49 mouse T lymphoma cells. Methods Enzymol. 1987;151:9-19. doi: 10.1016/s0076-6879(87)51005-9. No abstract available. PMID 3501530
- [Background] Farmer C, Fenu E, O'Flynn N, Guthrie B. Clinical assessment and management of multimorbidity: summary of NICE guidance. BMJ. 2016 Sep 21;354:i4843. doi: 10.1136/bmj.i4843. No abstract available. PMID 27655884
- [Background] Liu J, Liu P, Ma Z, Mou J, Wang Z, Sun D, Cheng J, Zhang D, Xiao J. The effects of aging on the profile of the cervical spine. Medicine (Baltimore). 2019 Feb;98(7):e14425. doi: 10.1097/MD.0000000000014425. PMID 30762749
- [Derived] Li YC, Chen KH, Li CY, Lu YJ. The outcome of injured cervical spinal cord with uncontrolled swelling under duraplasty: protocol of the ISCUD randomized controlled trial. Trials. 2025 Dec 2;26(1):559. doi: 10.1186/s13063-025-09288-6. PMID 41331929